CLINICAL TRIAL: NCT04085497
Title: Efficacy of Kinesio Tape in the Treatment of Medial Plica Syndrome - A Prospective Study
Brief Title: Kinesio Tape in the Treatment of Medial Plica Syndrome
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Istanbul Bilgi University (Other)
Responsible Party: Principal Investigator, TOMRIS DUYMAZ, Principal Investigator, Istanbul Bilgi University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MPS
Record Dates: First submitted 2019-09-09; First posted 2019-09-11 (Actual); Last update posted 2019-09-13 (Actual); Status verified 2019-09

CONDITIONS: Medial Plica Syndrome
Keywords: Medial Plica Syndrome; Kinesio Tape
MeSH Terms: interventions — Therapeutics

STUDY DESIGN:
Intervention Model Description: The patients were divided into two groups, each comprising 40 patients. KT and exercise were given to the patients in the first group, and only exercise was given to the patients in the second group. The inclusion criteria included patients between the ages of 20 and 55 who were diagnosed as MPS by MPP test and MRI imaging and did not develop cartilage damage. Patients with meniscal tear, chondral injury or instability of the knee were excluded.
Who Masked: Investigator
Masking Description: Single
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment (Experimental): KT was applied once a week, 6 times in total. Exercises were performed for all patients for 5 weeks 5 days a week, 3 sets 15 repetitions each day.
  Interventions: Other: Treatment
- Group 2 (Placebo Comparator): The exercise program included quadriceps set exercise, straight leg lifting, mini squat, stretching to hamstring and gastrosoleus muscle groups.
  Interventions: Other: Treatment

INTERVENTIONS:
Other: Treatment — KT application: KT application includes 2 stages. The banding in the first step is directed to the patellar tendon in order to absorb the load of the knee. The second step is directed directly on the medial plica to benefit from its analgesic effect. For the first step, an I-band is measured from the top of the patella to the tuberositas tibia. I-band is 6 cm wide and 5 mm thick. This I-band is cut into Y-band. First, the part of the band above the patella is pasted with 10% tension. Then the patient's knee is flexed to maximum flexion and the tails of the band are pasted around the patella with 0% tension. The tails of the band are combined together on the tuberositas and completed. For the second step, 4 I-bands 8 cm long and 1.5 cm wide are prepared. The middle of the I-bands is attached to the medial plica with a 0% tension, giving a star shape.

SUMMARY:
The aim of this study was to investigate the efficacy of kinesio tape (KT) on pain severity, pain threshold, lower extremity functional muscle strength and dynamic balance, functional status, and quality of life in patients with Medial Plica Syndrome (MPS).

DETAILED DESCRIPTION:
This randomized prospective controlled trial was designed, conducted and reported in accordance with the standards of the CONSORT (Consolidated Standards of Reporting Trials) statement. The approval of the Istanbul Bilgi University Clinical Investigations Ethics Committee was obtained, and the enrolled subjects signed a free and informed consent form.

Trial design KT was applied once a week, 6 times in total. Exercises were performed for all patients for 5 weeks 5 days a week, 3 sets 15 repetitions each day. The exercise program included quadriceps set exercise, straight leg lifting, mini squat, stretching to hamstring and gastrosoleus muscle groups.

Intervention KT application: KT application includes 2 stages. The banding in the first step is directed to the patellar tendon in order to absorb the load of the knee. The second step is directed directly on the medial plica to benefit from its analgesic effect. For the first step, an I-band is measured from the top of the patella to the tuberositas tibia. I-band is 6 cm wide and 5 mm thick. This I-band is cut into Y-band. First, the part of the band above the patella is pasted with 10% tension. Then the patient's knee is flexed to maximum flexion and the tails of the band are pasted around the patella with 0% tension. The tails of the band are combined together on the tuberositas and completed. For the second step, 4 I-bands 8 cm long and 1.5 cm wide are prepared. The middle of the I-bands is attached to the medial plica with a 0% tension, giving a star shape.

Participants The study was included 80 patients with diagnosed as MPS in the Orthopedics and Traumatology outpatient clinic of Bağcılar Training and Research Hospital. MPS was diagnosed by MRI imaging in patients with pain and MPP test in the patella anteromedial. The patients were divided into two groups, each comprising 50 patients. KT and exercise were given to the patients in the first group, and only exercise was given to the patients in the second group. The inclusion criteria included patients between the ages of 20 and 55 who were diagnosed as MPS by MPP test and MRI imaging and did not develop cartilage damage. Patients with meniscal tear, chondral injury or instability of the knee were excluded.

Outcome measurements Measurements were performed twice before and after the treatment for all patients. Pain threshold with digital algometer, pain severity with visual analog scale (VAS), disability level with Lysholm Knee Scoring Scale, functional strength and dynamic balance of lower extremity with stairs up and down test, quality of life with Nottingham Health Profile (NHP) were evaluated before and after treatment.

ELIGIBILITY:
Inclusion Criteria:

* Patients between the ages of 20 and 55
* Diagnosed as medial plica syndrome by MPP test and MRI imaging
* Did not develop cartilage damage

Exclusion Criteria:

* Patients with meniscal tear, chondral injury or instability of the knee

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 80 (Estimated)
Dates: Start 2019-01-02 (Actual); Primary Completion 2019-05-10 (Actual); Study Completion 2019-10-01 (Estimated)

PRIMARY OUTCOMES:
Pain threshold | 1 minute
  Algometer is a tool that measures pressure pain threshold and pain tolerance in quantitative sensory tests

SECONDARY OUTCOMES:
Pain severity: score | 1 minutes
  Participants were told how to do it and were asked to give a score between 0-100
Disability scale | 5 minutes
  The Lysholm Knee Scoring scale is a scale used in all knee injuries. 8 parameters (limp, using cane or crutches, locking sensation in the knee, giving way sensation from the knee, pain, swelling, climbing stairs, squatting) are evaluated.When calculating the score, the most appropriate option is selected in each parameter and the total score is found by adding the scores obtained from the whole parameter. Lysholm knee score; ≥95 points are rated as 'excellent', 84-94 points as 'good', 65-83 points as 'moderate', ≤64 points as 'bad'.
Nottingham Health Profile | 8 minutes
  The Nottingham Health Profile (NHP) was used to determine quality of life of the participants. This scale consists of 38 items formed as yes-no questions that cover 6 subscales of the quality of life. These six subscales are sleep (5 item), energy level (3 item), emotional status (9 item), social isolation (5 item), physical mobility (8 item) and pain (8 item). Each section is scored from 0-100. 0 indicates the best health status, 100 indicates the worst health status.

CONTACTS AND LOCATIONS:
Overall Officials: Tomri̇s Duymaz, Principal Investigator — Istanbul Bilgi University
Locations (1):
- Istanbul Bilgi University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No